CLINICAL TRIAL: NCT04655898
Title: A Phase 1, Single-Center, Open-label Study to Evaluate the Metabolism and Exception of [14C]-CC-90001 in Healthy Male Subjects
Brief Title: Metabolism and Excretion of [14C]CC-90001 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90001-CP-007; U1111-1261-4819 (Registry Identifier: WHO)
Record Dates: First submitted 2020-12-03; First posted 2020-12-07 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteer
Keywords: Mass balance; Males; Healthy volunteers; CC-90001; [14C]CC-90001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of [14C]CC-90001 (Experimental): A single oral dose of [14C]CC-90001, containing approximately 100 μCi of radioactivity, will be administered on Day1 under fasted conditions.
  Interventions: Drug: [14C]CC-90001

INTERVENTIONS:
Drug: [14C]CC-90001 — Oral

SUMMARY:
This is a clinical pharmacology study to characterize the biotransformation and excretion of [14C]CC-90001 and to evaluate the safety and tolerability of [14C]CC-90001 following a single oral dose of [14C]CC-90001 in healthy male subjects. Approximately 8 subjects will be enrolled into the study with a goal of 6 subjects being eligible for analysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥18 and ≤55 years of age, from any race, at the time of signing the informed consent form (ICF).
2. Subject is a male.
3. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
4. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
5. Subject is in good health, as determined by the Investigator based on a physical examinations and laboratory testing at screening or at check-in.
6. Must practice true abstinence or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of childbearing potential (FCBP) on the day of taking the single dose of study drug and for at least 90 days after taking the single dose of study drug. This also applies to those subjects who have had a successful vasectomy.
7. Subject has a body mass index (BMI) ≥ 18 and ≤ 33kg/m2 at screening.
8. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 160mmHg, supine diastolic BP ≥ 50 and ≤ 100 mmHg, and pulse rate ≥ 40 and ≤ 90bpm at screening and check-in.
9. Subject has screening laboratory test results within the reference range or, if outside the reference range, documented to be not clinically significant by the Investigator.
10. Subject has a normal or clinically acceptable 12-lead electrocardiogram (ECG), with a QT interval corrected using Fredericia formula (QTcF) value ≤ 450 msec, at screening and check-in

Exclusion Criteria:

1. Subject has any significant medical condition, laboratory observation, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including a laboratory test result which places the subject at unacceptable risk if he were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject was exposed to an investigational drug (new chemical entity) within 30days prior to dosing, or 5half-lives of that investigational drug, if known (whichever is longer).
5. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 14 days or 5 half-lives of that medication, whichever is longer, prior to dosing.
6. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 7days prior to dosing.
7. Subject has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30days prior to dosing. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP3A (http://medicine.iupui.edu/clinpharm/ddis/table.aspx). Please consult the medical monitor for any uncertainties with regard to potential CYP3A modulators.
8. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure or Gilbert's syndrome.

   a. Note: prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study. Please consult the medical monitor for uncertainties around the relevance of prior surgical procedures.
9. Has donated blood or plasma within 2weeks before dose administration to a blood bank or blood donation center.
10. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to dosing, or positive drug test reflecting consumption of drugs of abuse.
11. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years prior to dosing, or positive alcohol test.
12. Positive SARS-CoV-2 (severe acute respiratory syndrome coronavirus) test or signs/symptoms of COVID-19 (Coronavirus Disease 2019) infection.
13. Subject is known to have serum hepatitis or be a carrier of Hepatitis B virus (HBV) or Hepatitis C virus (HCV); or express hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
14. Smokers or users of other tobacco products (self-reported).
15. Subject has received immunization with a live or live attenuated vaccine within 1 months prior to dosing or is planning to receive immunization with a live or live attenuated vaccine for 1months following dosing.
16. Subjects who have participated in more than one other radiolabeled investigational drug study within 12 months prior to Check-in (Day-1).

    a. Note: The previous radiolabeled investigational drug must have been received more than 6 months prior to check-in (Day-1) and the total planned exposure from this current study and the previous study must be within the recommended levels considered safe, per US code of federal regulations (CFR) governing Protection of Human Subjects; radioactive drugs for certain research uses (ie, less than 5000 mrem whole body annual exposure; 21CFR361.1).
17. Subject was exposed to serial X-ray or computed tomography scans, barium meal, or employment in a job requiring radiation exposure monitoring within 12 months prior to Day-1.
18. History of less than 1 to 2 bowel movements per day.
19. Subject is part of the study site personnel or a family member of the study site staff.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Total [14C]-RA | Up to approximately 216 hours post dose
  Total [14C]-Radioactivity (RA) in whole blood, plasma, urine, and feces) will be measured via Liquid scintillation counting (LSC)
Pharmacokinetics - Cumulative excretion of total [14C]-RA | Up to approximately 13 days
  The total recovery of radioactivity will be computed as the sum of the cumulative excretion (as % dose) in urine and feces
Pharmacokinetics - Total [14C]-RA whole blood-to-plasma ratios | Up to approximately 216 hours post
  Total [14C]-RA in whole blood and plasma will be converted to ngEq/mL concentration of [14C]CC-90001 based on specific activity of the dose. Equivalent concentration-time profiles will be determined.
Pharmacokinetics - metabolite profiling in plasma | Up to approximately 216 hours post
  The RA will be determined for CC-90001 and any identified metabolites in plasma. Metabolite profiling may use pooled time points.
Pharmacokinetics - metabolite profiling in urine and feces | Up to approximately 13 days
  Percentage of the administered dose, and the RA, will be determined for CC-90001 and any identified metabolites in urine and feces. Metabolite profiling may use pooled collection intervals.
Pharmacokinetics - Cmax | Up to approximately 216 hours post
  Observed maximum concentration of [14C]CC-90001 and for metabolites with sufficient measurable concentration
Pharmacokinetics - AUC | Up to approximately 216 hours post
  Area under the concentration-time curve of [14C]CC-90001 and for metabolites with sufficient measureable concentration
Pharmacokinetics - Tmax | Up to approximately 216 hours post
  Time to Cmax of [14C]CC-90001 and for metabolites with sufficient measureable concentration
Pharmacokinetics - t1/2 | Up to approximately 216 hours post
  Terminal elimination half-life of [14C]CC-90001 and for metabolites with sufficient measureable concentration

SECONDARY OUTCOMES:
Number of treatment-emergent adverse event related to CC-90001 | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/